CLINICAL TRIAL: NCT00506493
Title: Medtronic Concomitant Utilization of Radio Frequency Energy for Atrial Fibrillation (CURE-AF)/Persistent Study
Brief Title: Medtronic Concomitant Utilization of Radio Frequency for Atrial Fibrillation CURE-AF/Persistent
Acronym: CURE-AF/Perst
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Cardiac Surgery (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CURE-AF/Persistent
Record Dates: First submitted 2007-07-22; First posted 2007-07-25 (Estimated); Results first posted 2013-10-16 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation Surgical RF Ablation; Perisistent Atrial Fibrillation; Surgical Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cardioblate Surgical Ablation System — This investigation is a prospective, nonrandomized multicenter clinical trial evaluating the outcome of patients with AF requiring concomitant open heart surgery plus the Cardioblate Surgical Ablation System using the modified Maze III procedure. The trial population includes patients requiring valve replacements or repairs, atrial septal defect (ASD) repairs, patent foramen ovale (PFO) closure or coronary artery bypass grafts (CABG) procedures.
Procedure: Surgical RF Ablation — This investigation is a prospective, nonrandomized multicenter clinical trial evaluating the outcome of patients with AF requiring concomitant open heart surgery plus the Cardioblate Surgical Ablation System using the modified Maze III procedure. The trial population includes patients requiring valve replacements or repairs, atrial septal defect (ASD) repairs, patent foramen ovale (PFO) closure or coronary artery bypass grafts (CABG) procedures.

SUMMARY:
This investigation is a prospective, nonrandomized multicenter clinical trial evaluating the outcome of patients with atrial fibrillation (AF) requiring concomitant open heart surgery plus the Cardioblate Surgical Ablation System using the modified Maze III procedure. The trial population includes patients requiring valve replacements or repairs, atrial septal defect (ASD) repairs, patent foramen ovale (PFO) closure or coronary artery bypass graft (CABG) procedures. The study objectives are to demonstrate that the Medtronic Cardioblate Surgical Ablation System can safely and effectively treat persistent AF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a documented history of persistent AF as defined by the ACC/AHA/ESC Guidelines: Characterized as episodes of non-self-terminating atrial fibrillation that usually lasts more than 7 days.
2. Concomitant indication (other than AF) for open-heart surgery for one or more of the following:

   * Mitral valve repair or replacement
   * Aortic valve repair or replacement
   * Tricuspid valve repair or replacement
   * Atrial septal defect (ASD) repair
   * Patent foramen ovale (PFO) closure
   * Coronary artery bypass procedures
3. Greater than or equal to 18 years of age
4. Able and willing to comply with study requirements by signing a consent form
5. Must be able to take the anticoagulant warfarin (Coumadin)

Exclusion Criteria:

1. Wolff-Parkinson-White syndrome
2. NYHA Class = IV
3. Left ventricular ejection fraction ≤ 30%
4. Need for emergent cardiac surgery (i.e. cardiogenic shock)
5. Previous atrial ablation for AF, AV-nodal ablation, or surgical Maze procedure
6. Contraindication for anticoagulation therapy
7. Left atrial diameter > 7.0 cm
8. Preoperative need for an intra-aortic balloon pump or intravenous inotropes
9. Renal failure requiring dialysis or hepatic failure
10. Life expectancy of less than one year
11. Pregnancy or desire to be pregnant within 12 months of the study treatment.
12. Current diagnosis of active systemic infection
13. Documented MI 6 weeks prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-09; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thoralf Sundt, MD, Principal Investigator — The Mayo Clinic- Rochester
Locations (15):
- United States (15):
  - Southwest Heart and Lung, Phoenix, Arizona
  - East Bay Cardiovascular & Thoracic Associates, Concord, California
  - University of Southern California, Los Angeles, California
  - Eisenhower Medical Center, Palm Springs, California
  - Cardiac Surgical Associates of Florida, St. Petersburg, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Mayo/St. Mary's Hospital, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Lenox Hill Hospital, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Inova Fairfax, Falls Church, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 90 subjects were consented into the study, of which 75 subjects received study treatment at 13 of the 15 investigational centers in the United States. The first subject was enrolled on September 18, 2007 and last patient enrolled on October 27, 2010.
Pre-assignment Details: No additional wash out, run-in, or transition was utilized during this study. A subject was considered enrolled once treatment occurred.
Groups:
- Cardioblate Surgical Ablation System: 75 subjects were enrolled and treated. 64 subjects completed the study through the 9 month follow-up. 6 subjects died and 5 subjects withdrew from the study.
Period: Overall Study
Arm/Group | Cardioblate Surgical Ablation System
Started | 75
Completed | 64
Not Completed | 11
Not completed — Death | 6
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Groups:
- Study Completion Cohort: 75 subjects were enrolled and treated. 64 subjects completed the study through the 9 month follow-up. 6 subjects died and 5 subjects withdrew from the study.
Arm/Group | Study Completion Cohort
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint: The Percent of Patients Off Class I or III Antiarrhythmic Drugs and Out of AF as Determined by 24 Hour Holter Recording at 9 Months
Description: Subject's cardiac rhythm was assessed by wearing a Holter Monitor for 24 hours
Time Frame: 9 months
Population: 75 subjects were enrolled, 14 subjects had no Holter assessment performed- 6 subjects died, 5 subjects withdrew participation, and 3 subjects completed endpoint follow-up without analyzable Holter data.
Measure: Number; unit: percentage of subjects
Groups:
- Cardioblate Surgical Ablation System: All subjects enrolled who underwent surgical ablation with the Cardioblate Surgical Ablation system and completed a Holter assessment at 9 month follow-up
Arm/Group | Cardioblate Surgical Ablation System
Number analyzed (Participants) | 61
percentage of subjects | 42.6
Statistical Analysis 1: Comparison: Cardioblate Surgical Ablation System; The specific test hypothesis is as follows: H0: ptest ≤ 22.1% Ha: ptest > 22.1%; Test type: Superiority or Other; p < 0.01, Fisher Exact — The percent of patients off Class I and III AADs and successfully converted out of AF following treatment (ptest) will exceed the percent of patients off Class I and III AADs and convereted out of AF, as reported in literature (pcontrol=22.1%); Binomial Proportions = 42.6, 97.5% CI 1-sided [lower limit 30.0], Standard Error of Mean 6.3

2. Primary Outcome: Safety Endpoint: Composite Acute Major Adverse Event Rate, Within 30 Days Post-procedure or Hospital Discharge
Description: Major Adverse Events were defined to include: mediastinitis, death, myocardial infarction, stroke, transient ischemic attacks (TIA), pulmonary embolism, peripheral arterial embolism, and esophageal injury.
Time Frame: 30 days post procedure or hospital discharge
Measure: Number; unit: percentage of subjects
Groups:
- Cardioblate Surgical Ablation System: All subjects who underwent surgical ablation with the Cardioblate Surgical Ablation System.
Arm/Group | Cardioblate Surgical Ablation System
Number analyzed (Participants) | 75
percentage of subjects | 6.7 [lower limit 0]
Statistical Analysis 1: Comparison: Cardioblate Surgical Ablation System; Test type: Superiority or Other; p < 0.0001, Fisher Exact; binomial proportions = 6.7, 97.5% CI 1-sided [upper limit 14.9]

3. Secondary Outcome: Efficacy Endpoints: The Percent of Patients Out of AF, Regardless of Antiarrhythmic Drug Status, as Determined by a 24 Hour Holter Recording at 9 Months
Time Frame: 9 months
Measure: Number; unit: percentage of subjects
Groups:
- Cardioblate Surgical Ablation System: 75 subjects were enrolled and treated with the Cardioblate Surgical Ablation System.. 64 subjects completed the study through the 9 month follow-up. 6 subjects died and 5 subjects withdrew from the study.
Arm/Group | Cardioblate Surgical Ablation System
Number analyzed (Participants) | 61
percentage of subjects | 67.2

4. Secondary Outcome: Safety Endpoints: Composite 9-month Major Adverse Event Rate, Post-procedure
Description: as for outcome 2
Time Frame: 9 months
Measure: Number; unit: percentage of subjects
Arm/Group | Cardioblate Surgical Ablation System
Number analyzed (Participants) | 70
percentage of subjects | 11.4

ADVERSE EVENTS:
Time Frame: Adverse events reported from treatment through 9 month follow-up.
Description: This study was overseen by a Data Safety Monitoring Board (DSMB) and a Clinical Events Committee (CEC). The DSMB reviewed the data and made recommendations regarding any safety concerns and also assessed the data from a risk/benefit perspective. The CEC reviewed and adjudicated MAEs and serious adverse events (SAEs).
Arm/Group | Study Completion Cohort
Serious Adverse Events (participants affected / at risk) | 45/75
Other Adverse Events (participants affected / at risk) | 59/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Completion Cohort (N=75)
Endocarditis (Infections and infestations) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 1 (1)
Hemodynamic Instability (Cardiac disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 3 (3)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection/Sepsis (Infections and infestations) | 5 (5)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 20 (21)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrioventricular Third Degree AV Heart Block (Cardiac disorders) | 2 (2)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Insufficiency/Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Renal Insufficiency/Failure: Dialysis Required (Renal and urinary disorders) | 5 (5)
Renal Insufficiency/Failure: No Dialysis Required (Renal and urinary disorders) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhythms with Potentially Deleterious Hemodynamic Consequences Requiring Intervention (Cardiac disorders) | 5 (7)
Shock (Cardiac disorders) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 3 (3)
Cardiac Tamponade (Cardiac disorders) | 3 (3)
Congestive Heart Failure (Cardiac disorders) | 8 (8)
Angina Presenting as SOB (Cardiac disorders) | 1 (1)
Ascites with Paracentesis (Hepatobiliary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial Fibrillation/Atrial Flutter/Bradycardia (Cardiac disorders) | 2 (2)
Atrial tachycardia with dyspnea on exertion (Cardiac disorders) | 1 (1)
Chest tube site wound (Skin and subcutaneous tissue disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Flu (General disorders) | 1 (1)
Herniated lumbar disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Liver Failure (Endocrine disorders) | 1 (1)
Liver Shock (Endocrine disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Pain/discomfort on pacer site, right subclavian area (Musculoskeletal and connective tissue disorders) | 1 (1)
Rectal Bleeding (Renal and urinary disorders) | 1 (1)
Sternal Dehiscence (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper Extremity Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Completion Cohort (N=75)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Hemodynamic Instability (Cardiac disorders) | 7 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Renal Insufficiency/Failure: No Dialysis Required (Renal and urinary disorders) | 9 (9)

LIMITATIONS AND CAVEATS:
* Slow/delayed enrollment
* Medical management of subjects by non-investigators leading to medication washout protocol deviations
* Missing endpoint data (attrition) due to cohort demographics (old age, dementia, relocation, etc.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less